CLINICAL TRIAL: NCT05859178
Title: Exercise Training to Improve Nerve Regeneration and Function in Patients With Brachial Plexus Injury Following Nerve Transfer - a Randomized Controlled Clinical Trial
Brief Title: Exercise Training for Brachial Plexus Injury Following Nerve Transfer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other); Glenrose Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00128785
Record Dates: First submitted 2023-04-05; First posted 2023-05-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brachial Plexus Injury

STUDY DESIGN:
Intervention Model Description: Participants assigned to the exercise group will perform strengthening exercise. Those assigned to the control group will carry out stretch exercise that is not known to have any effect on nerve regeneration.
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessor will not be involved in treatment delivery. Participants in the control group will carry out sham exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Each participant in the exercise group will undergo hand grip exercise for 30 minutes a day, 5 days a week for a total of 12 weeks. To activate the ulnar nerve innervated muscles, the exercise will be done using an electronic hand grip device with adjustable resistance individualized to the strength of each participant.
  Interventions: Other: Exercise group
- Control group (Experimental): Participants will carry out a stretch exercise routine that is not known to have any effect on nerve regeneration.
  Interventions: Other: Exercise group

INTERVENTIONS:
Other: Exercise group — Along with nerve transfer surgery, individuals in the exercise group will undergo handgrip exercise for 30 minutes a day, 5 days a week for a total of 12 weeks.

SUMMARY:
Although peripheral nerve is capable of regrowth following injury, at only 1 mm/day, the slow rate represents a major barrier. Apart from rapid deterioration of the environment supportive of growth, denervated muscles become atrophic and bones osteoporotic. To successfully restore function, in addition to speeding up the nerve regeneration rate, treatments that can also restore muscle and bone mass are essential. Recently, in animal studies, the investigators showed that in addition to accelerating the speed of nerve regeneration, exercise training can also be used to restore muscle bulk and bone density. While promising, given the inter-species differences, the clinical utilities of this treatment need to be directly tested in humans. This will be done using a randomized controlled study design on patients with brachial plexus injury.

DETAILED DESCRIPTION:
Peripheral nerve injury is common, affecting 3% of patients with limb trauma seen in the emergency department. Of those, young males who are active in the work force are most frequently inflicted. The functional loss does not only carry a huge personal burden but is also associated with substantial healthcare and socioeconomic costs. Indeed, based on data from the National Inpatient Sample in the US, estimated direct healthcare costs for patients who sustained upper limb nerve injury is over $1.2B per year. Although in previous studies the investigators found that conditioning electrical stimulation, a form of activity dependent therapy, enhances nerve regeneration following injury, it did not improve bone density. Therefore, alternative treatments capable of promoting bone formation, restoring muscle bulk and increasing nerve regeneration are needed.

Based on recent discoveries in animal studies, the goal of this randomized controlled clinical trial is to test the hypothesis that exercise training can accelerate nerve regeneration and significantly increase muscle bulk and bone density compared to surgery alone in patients with brachial plexus injury.

To test this hypothesis, patients with brachial plexus injury involving the musculocutaneous nerve will be randomized to the exercise or control group following nerve transfer surgery. This will be done using a redundant branch of the ulnar nerve to reinnervate the biceps muscle. To evaluate the treatment efficacy, compound muscle action potential of the biceps muscle will be used as the primary outcome measure to quantify reinnervation. The following anatomic and functional measures will be used as secondary outcome measures: i) muscle bulk of the biceps using MRI; ii) bone density of the humerus using dual-energy x-ray absorptiometry (DEXA) imaging; iii) quantitative force measurement for elbow flexion; iv) the Disability of Arm, Shoulder and Hand (DASH) instrument to assess disability, and v) the Canadian Occupational Performance Measure for limitations in participation.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18-60
* electrodiagnostically confirmed brachial plexus injury affecting the musculocutaneous nerve
* able to consent for participation.

Exclusion Criteria:

• individuals with additional neurological or musculoskeletal conditions that would affect elbow and hand function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Motor nerve conduction study | Baseline, 3, 6 and 9 months post surgery
  compound muscle action potential of the biceps muscle. Range: 0-7 mV. Higher scores signify better nerve regeneration

SECONDARY OUTCOMES:
magnetic resonance imaging (MRI) | Baseline, 3, 6 and 9 months post surgery
  muscle bulk of the biceps. Measure in cubic cm. Higher score signifies better nerve regeneration.
dual energy x-rays absorptiometry (DEXA) | Baseline, 3, 6 and 9 months post surgery
  bone density - humerus (g/sq. m). Higher scores denote better outcome
quantitative force measurement for elbow flexion using dynamometer DASH Questionnaire | Baseline, 3, 6 and 9 months post surgery
  to assess impairment (N). Higher scores denote better outcome
Canadian Occupational Performance Measure (COPM) | Baseline, 3, 6 and 9 months post surgery
  to assess handicap and participation (Range 1-5). Higher scores denote better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No